CLINICAL TRIAL: NCT03052153
Title: Intraoperative Echocardiographic Evaluation of Pulmonary Vein Velocities and Outcomes in Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Amar Bhatt, Attending Physician, Ohio State University
Other Study IDs: 2016H0435
Record Dates: First submitted 2017-01-07; First posted 2017-02-14 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Lung Transplant Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Transplant Surgery: Subjects included in the study will have undergone a single or bilateral lung transplant surgery at The Ohio State University Wexner Medical Center between 01 JAN 2014 and 18 NOV 2016. No investigational intervention performed for this study.
  Interventions: Other: No investigational intervention performed for this study

INTERVENTIONS:
Other: No investigational intervention performed for this study — No investigational intervention for the purpose of this study was performed; data collected is retrospective data previously collected for non-research purposes.

SUMMARY:
This study will evaluate if an association exists between levels of blood flow through the pulmonary veins and the incidence of graft dysfunction post operatively.

DETAILED DESCRIPTION:
Lung transplantation surgery can be fraught with a multitude of early as well as delayed complications leading to increased morbidity and mortality. During lung transplant surgery, trans-esophageal echocardiography (TEE) is routinely used to identify cardiac anatomy and measure blood flow through the pulmonary veins. This blood flow is assessed both before and after the lung has been transplanted. Blood flow through these small caliber vessels can be impacted by many variables with a resulting reduction in blood circulating to the lung, although currently there is no agreement on an acceptable level of flow. This study will look at retrospective data from lung transplant surgeries undertaken at this institution since Jan 1st 2014 until November 18th 2016 with the goal of determining if an association exists between levels of blood flow through the pulmonary veins and the incidence of graft dysfunction post operatively.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients ≥ 18 years of age
2. Having undergone single or bilateral lung transplantation surgery at Ohio State University Wexner Medical Center between January 1st 2014 and November 18th 2016

Exclusion Criteria:

1. Patients ≤ 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all surgical patients 18 years of age and older who underwent single or bilateral lung transplantation surgery during the period January 1st 2014 to November 18 2016 at Ohio State University Wexner Medical Center. Database screening for patient inclusion in retrospective analysis will be performed by designated personnel from the Anesthesiology Department or co-investigators entitled to work with patients' electronic data.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
incidence of graft dysfunction | at 30 days post-transplant
  To describe the relationship between intra-operative pulmonary vein systolic velocities and the incidence of graft dysfunction as defined by the International Society for Heart and Lung Transplantation (ISHLT).
grade of graft dysfunction | at 30 days post-transplant
  To describe the relationship between intra-operative pulmonary vein systolic velocities and grade of graft dysfunction as defined by the International Society for Heart and Lung Transplantation (ISHLT).

SECONDARY OUTCOMES:
All-cause mortality | at 30 days post-transplant
  To measure and report all-cause mortality at 30 days post-transplant.
Hospital Length of Stay | From hospital admission to discharge up to one year.
  To report subjects hospital length of stay for up to one year.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Bhatt, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No